CLINICAL TRIAL: NCT02217930
Title: A Randomized, Double-Blind, Double-Dummy, Placebo- and Positive- Controlled, Crossover Study to Evaluate the Effect Of WCK 2349 on the QT/QTc Interval in Health Volunteers
Brief Title: Study to Evaluate the Effect Of WCK 2349 on the QT/QTc Interval in Health Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: W-2349-101
Record Dates: First submitted 2014-07-31; First posted 2014-08-15 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Qt Interval, Variation in
Keywords: TQT
MeSH Terms: interventions — levonadifloxacin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo matched to WCK 2349, oral tablet(s)
  Placebo matched to moxifloxacin overencapsulated tablet
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): Moxifloxacin 400 mg positive control (overencapsulated tablet)
  Interventions: Drug: Moxifloxacin
- WCK 2349 (Experimental): WCK 2349 supratherapeutic dose determined in Part 1, oral tablet(s)
  Interventions: Drug: WCK 2349

INTERVENTIONS:
Drug: WCK 2349
  Arms: WCK 2349
Drug: Placebo
  Arms: Placebo
Drug: Moxifloxacin
  Arms: Moxifloxacin

SUMMARY:
The study designed to determine the effect induced by WCK 2349 on the QT interval.

The study will be conducted in two parts: 1) to determine the supratherapeutic dose; and 2) to assess the safety of high doses of single-dose administration of WCK 2349 on the QT interval.

DETAILED DESCRIPTION:
Part 1 of this study will determine the supratherapeutic dose to be used in Part 2. Part 1will enroll 8 subjects at each of 4 dose levels (up to 32 subjects). Cohorts will be staggered so that appropriate safety monitoring and follow-up can be performed for each subject at each dose level.

Safety monitoring will be based upon review of AEs, ECGs and clinical laboratory test results prior to escalation to the next dose level.

At the first dose level, 6 subjects will be randomly assigned to receive a single dose of WCK 2349 at 1800 mg and 2 subjects will be randomly assigned to placebo. If this dose is tolerated by subjects, and safety data allows, the next group will be initiated in the same fashion at a dose of 2200 mg. If this dose is tolerated by subjects, and safety data allows, the next group will be initiated in the same fashion at a dose of 2600 mg. If this dose is tolerated by subjects, and safety data allows, the next group will be initiated in the same fashion at a dose of 3000 mg. Based upon safety data, the highest safely tolerated dose in Part 1 will be utilized as the supratherapeutic dose in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 18 and 55 years of age,inclusive, with a body mass index ≥18 to ≤33 kg/m2.
* Female subjects must be at least 2 years postmenopausal,surgically sterile, or practicing 2 highly effective methods of birth control (determined by the investigator or designee; one of the methods must be a barrier technique), not pregnant or lactating, and have a negative serum pregnancy test before enrolling in the study.
* Male or female subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from Screening until 30 days after the last dose of study drug.
* Stable health based on no clinically significant findings on the medical history, physical examination, or clinical laboratory test results (as determined and documented by the investigator).
* Willing to comply with all study activities and procedures and provides written informed consent prior to any study procedures.

Exclusion Criteria:

1. An uninterpretable or abnormal screening electrocardiogram (ECG) indicating a second- or third-degree atrioventricular block, or one or more of the following: QRS interval >110 milliseconds (msec); QT interval corrected by Fridericia's formula (QTcF) >430 msec (males) and >450 msec (females); PR interval >200 msec; heart rate (HR) <45 bpm; or any rhythm other than sinus rhythm that is interpreted by the investigator to be clinically significant.
2. History of risk factors for torsades de pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments including hypokalemia, hypercalcemia, or hypomagnesemia. Subjects will also be excluded if there is a family history of long QT syndrome or Brugada syndrome.
3. A sustained supine systolic blood pressure >150 mm Hg or <90 mm Hg or a supine diastolic blood pressure >95 mm Hg or <50 mm Hg at Screening or Check-in (Day -1). Blood pressure may be retested once in the supine position. The blood pressure abnormality is considered sustained if either the systolic or the diastolic pressure values are outside the stated limits after 2 assessments, and the subject may not be randomized.
4. A resting HR of <40 beats per minute or >100 beats per minute when vital signs are measured at Screening or Check-in (Day -1).
5. Unstable cardiovascular disease, including recent myocardial infarction or cardiac arrhythmia.
6. Uncontrolled hypertension, asthma, unstable diabetes (type I or type II), thyroid disease, seizures, myasthenia gravis, or any other neuromuscular disorder.
7. Women who are pregnant (or planning to become pregnant within the next 6 months) or currently breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in QTc interval | Baseline and 48 hours

SECONDARY OUTCOMES:
Highest dose of WCK 2349 tolerated | Baseline and 48 hours
Number of Adverse Events | Baseline and 7 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical Research Inc.
Locations (1):
- Phase 1 unit : Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States